CLINICAL TRIAL: NCT01215279
Title: A 4-week, Double-Blind, Placebo-Controlled, Randomised, Parallel Group, Multi-Centre, Phase IIa Study to Investigate the Tolerability and Safety of 100 mg Oral AZD2423 in Patients With Moderate to Severe COPD
Brief Title: AZD2423 Safety and Tolerability Study in Patients With Moderate and Severe Chronic Obstructive Pulmonary Disease(COPD)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: D3320C00002
Record Dates: First submitted 2010-09-30; First posted 2010-10-06 (Estimated); Results first posted 2014-10-23 (Estimated); Last update posted 2014-10-23 (Estimated); Status verified 2014-10

CONDITIONS: Chronic Obstructive Pulmonary Disease; Lung Disease
Keywords: Respiratory disease; Chronic Obstructive Pulmonary Disease
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Lung Diseases; Respiration Disorders

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- AZD2423 (Experimental): AZD2423 Oral Treatment for 28 days
  Interventions: Drug: AZD2423
- Placebo (Placebo Comparator): Oral treatment for 28 days
  Interventions: Drug: Placebo to AZD2423

INTERVENTIONS:
Drug: AZD2423 — 100 mg oral treatment once daily for 28 days
  Arms: AZD2423
Drug: Placebo to AZD2423 — Oral treatment once daily for 28 days
  Arms: Placebo

SUMMARY:
The purpose of the study is to investigate the tolerability and safety of AZD2423 in Patients with chronic obstructive pulmonary disease.

ELIGIBILITY:
Inclusion Criteria:

* Male or female of non-child bearing potential. Only women of non-child bearing potential are included in the study i.e. women who are permanently or surgically sterilised or post menopausal.
* Between 40 and 80 years of age at Visit 1
* Clinical diagnosis of COPD (GOLD stage 2 or 3)
* FEV1/FVC <70% and FEV1 between 30 and 80% of the predicted normal post-bronchodilator (GOLD stage 2 or 3)
* Current or ex-smokers

Exclusion Criteria:

* Any clinically significant disease or disorder (including history of abnormal immune function) which, in the opinion of the Investigator, may either put the subject at risk or influence the way the drug works
* Any lung disease other than COPD, recent respiratory infections which have not resolved fully, active tuberculosis or at risk of reactivation of tuberculosis.
* Any abnormal findings in physical examination, blood or urine test results, vital signs or ECG at Visit 1 that may put the subject at risk during the study, affect their ability to take part or influence the results of the study
* Immunisation with a live vaccine within 3 months or other vaccination within 30 days before planned start of treatment
* Worsening of COPD symptoms within 4 weeks prior to start of study needing hospitalisation, oral steroids or antibiotics.

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 63 (Actual)
Dates: Start 2010-10; Primary Completion 2011-03 (Actual); Study Completion 2011-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Joanna Marks-Konczalik, MD, PhD, Study Director — AstraZeneca R&D
Locations (6):
- Bulgaria (2):
  - Research Site, Rousse
  - Research Site, Sofia
- Slovakia (4):
  - Research Site, Bratislava
  - Research Site, Košice
  - Research Site, Prešov
  - Research Site, Žilina

REFERENCES:
- See also: CSR-D3320C00002.pdf — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_MED_6111&studyid=207&filename=CSR-D3320C00002.pdf

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted at 11 centres in 2 countries: 5 in Bulgaria and 6 in Slovakia. The first patient was enrolled on 09 October 2010 and the last patient last visit was on 08 March 2011.
Groups:
- AZD2423 100 mg: Two 50 mg AZD2423 tablets, once daily for 28 days
- Placebo: Placebo to match AZD2423 50 mg tablets, once daily for 28 days
Period: Overall Study
Arm/Group | AZD2423 100 mg | Placebo
Started | 31 | 32
Completed | 31 | 32
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | AZD2423 100 mg | Placebo | Total
Number analyzed (Participants) | 31 | 32 | 63
Age, Continuous [Mean (Standard Deviation); unit: Years] | 62.5 (7.8) | 60.6 (7.2) | 61.6 (7.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 9 | 16
  Male | 24 | 23 | 47

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Clinically Significant Changes in Laboratory Variables Other Than Monocytes
Description: Number of all participants with clinically significant changes in laboratory variables, except monocyte, assessed at all the listed time points
Time Frame: Day 1, 1 week, 2 weeks, 3 weeks, 4 weeks and 5 weeks (follow-up)
Measure: Number; unit: Participants
Arm/Group | AZD2423 100 mg | Placebo
Number analyzed (Participants) | 31 | 32
Participants | 0 | 0

2. Primary Outcome: Number of Participants With Clinically Significant Changes in Vital Signs
Description: Number of participants with clinically significant changes in vital signs assessed at all the listed time points
Time Frame: Day 1, 1 week, 2 weeks, 3 weeks, 4 weeks and 5 weeks (follow-up)
Measure: Number; unit: Participants
Arm/Group | AZD2423 100 mg | Placebo
Number analyzed (Participants) | 31 | 32
Participants | 0 | 0

3. Primary Outcome: Number of Participants With Clinically Significant Changes in ECG Variables
Description: Number of participants with clinically significant changes in ECG variables assessed at all the listed time points
Time Frame: Day 1, 1 week, 2 weeks, 3 weeks, 4 weeks and 5 weeks (follow-up)
Measure: Number; unit: Participants
Arm/Group | AZD2423 100 mg | Placebo
Number analyzed (Participants) | 31 | 32
Participants | 0 | 0

4. Primary Outcome: Number of Participants With Clinically Significant Changes in Physical Examination
Description: Number of participants with clinically significant changes in physical examination assessed at all the listed time points
Time Frame: Day 1, 1 week, 2 weeks, 3 weeks, 4 weeks and 5 weeks (follow-up)
Measure: Number; unit: Participants
Arm/Group | AZD2423 100 mg | Placebo
Number analyzed (Participants) | 31 | 32
Participants | 0 | 0

5. Primary Outcome: Monocytes at Baseline
Description: Monocyte count in peripheral blood at baseline (Pre-dose, Day 1)
Time Frame: Day 1
Measure: Mean (Standard Deviation); unit: 10^9/L
Arm/Group | AZD2423 100 mg | Placebo
Number analyzed (Participants) | 30 | 28
10^9/L | 0.47 (0.136) | 0.43 (0.143)

6. Primary Outcome: Monocytes at End of Treatment
Description: Monocyte count in peripheral blood at end of treatment (4 weeks)
Time Frame: week 4
Measure: Mean (Standard Deviation); unit: 10^9/L
Arm/Group | AZD2423 100 mg | Placebo
Number analyzed (Participants) | 27 | 29
10^9/L | 0.43 (0.165) | 0.55 (0.178)

7. Primary Outcome: Monocytes at Follow-up
Description: Monocyte count in peripheral blood at follow-up (Week 5; 1 week after end of treatment)
Time Frame: week 5 (follow-up)
Measure: Mean (Standard Deviation); unit: 10^9/L
Arm/Group | AZD2423 100 mg | Placebo
Number analyzed (Participants) | 27 | 29
10^9/L | 0.50 (0.175) | 0.52 (0.196)

8. Secondary Outcome: Morning FEV1 at Baseline
Description: Measurements conducted by patient in morning upon rising, before intake of morning dose of investigational product but after clearing out mucus. Patients was to refrain from taking rescue medication prior to measurement if possible.
Time Frame: Average of 10 days of pre-treatment measurements (day -10 to -1)
Measure: Mean (Standard Deviation); unit: L
Arm/Group | AZD2423 100 mg | Placebo
Number analyzed (Participants) | 31 | 32
L | 1.3 (0.41) | 1.3 (0.44)

9. Secondary Outcome: Morning FEV1 During Last 7 Days of Treatment
Description: as for outcome 8
Time Frame: Average of the last 7 days of treatment (week 4)
Measure: Mean (Standard Deviation); unit: L
Arm/Group | AZD2423 100 mg | Placebo
Number analyzed (Participants) | 31 | 32
L | 1.3 (0.40) | 1.4 (0.52)

10. Secondary Outcome: Evening FEV1 at Baseline
Description: Measurement conducted by patient in evening.
Time Frame: Average of 10 days of pre-treatment measurements (day -10 to -1)
Measure: Mean (Standard Deviation); unit: L
Arm/Group | AZD2423 100 mg | Placebo
Number analyzed (Participants) | 31 | 32
L | 1.3 (0.43) | 1.4 (0.44)

11. Secondary Outcome: Evening FEV1 During Last 7 Days of Treatment
Description: Measurement conducted by patient in evening.
Time Frame: Average of the last 7 days of treatment (week 4)
Measure: Mean (Standard Deviation); unit: L
Arm/Group | AZD2423 100 mg | Placebo
Number analyzed (Participants) | 31 | 32
L | 1.2 (0.37) | 1.4 (0.51)

12. Secondary Outcome: Morning Peak Expiratory Flow (PEF) at Baseline
Description: as for outcome 8
Time Frame: Average of 10 days of pre-treatment measurements (day -10 to -1)
Measure: Mean (Standard Deviation); unit: L/minute
Arm/Group | AZD2423 100 mg | Placebo
Number analyzed (Participants) | 31 | 32
L/minute | 190.5 (74.73) | 185.5 (74.21)

13. Secondary Outcome: Morning PEF During Last 7 Days of Treatment
Description: as for outcome 8
Time Frame: Average of the last 7 days of treatment (week 4)
Measure: Mean (Standard Deviation); unit: L/minute
Arm/Group | AZD2423 100 mg | Placebo
Number analyzed (Participants) | 31 | 32
L/minute | 190.2 (77.24) | 196.4 (83.81)

14. Secondary Outcome: Evening PEF at Baseline
Description: Measurement conducted by patient in evening.
Time Frame: Average of 10 days of pre-treatment measurements (day -10 to -1)
Measure: Mean (Standard Deviation); unit: L/minute
Arm/Group | AZD2423 100 mg | Placebo
Number analyzed (Participants) | 31 | 32
L/minute | 192.3 (74.27) | 196.2 (79.92)

15. Secondary Outcome: Evening PEF During Last 7 Days of Treatment
Description: Measurement conducted by patient in evening.
Time Frame: Average of the last 7 days of treatment (week 4)
Measure: Mean (Standard Deviation); unit: L/minute
Arm/Group | AZD2423 100 mg | Placebo
Number analyzed (Participants) | 31 | 32
L/minute | 191.9 (82.17) | 204.7 (87.98)

16. Secondary Outcome: Exacerbations of Chronic Pulmonary Disease Tool (EXACT) Total Score at Baseline
Description: The EXACT Tool is a Patient Reported Outcome (PRO) measure; 14 items evaluated on 5- or 6-point scales; total score ranges from 0 to 100 (higher values indicate more severe exacerbation). Baseline is the mean value over the 7 days prior to randomisation.
Time Frame: Average of 7 days of pre-treatment measurements (day -7 to -1)
Measure: Mean (Standard Deviation); unit: Units on scale, 0-100
Arm/Group | AZD2423 100 mg | Placebo
Number analyzed (Participants) | 31 | 32
Units on scale, 0-100 | 44.4 (6.99) | 45.7 (8.49)

17. Secondary Outcome: EXACT Total Score During Last 7 Days of Treatment
Description: The EXACT Tool is a Patient Reported Outcome (PRO) measure; 14 items evaluated on 5- or 6-point scales; total score ranges from 0 to 100 (higher values indicate more severe exacerbation).
Time Frame: Average of the last 7 days of treatment (week 4)
Measure: Mean (Standard Deviation); unit: Units on scale, 0-100
Arm/Group | AZD2423 100 mg | Placebo
Number analyzed (Participants) | 31 | 32
Units on scale, 0-100 | 43.8 (7.78) | 44.6 (9.84)

18. Secondary Outcome: Breathlessness, Cough and Sputum Scale (BCSS) (Evening) Total Score at Baseline
Description: The BCSS scale includes one question for each of the symptoms of breathlessness, cough, and sputum. The total BCSS score ranges from 0 to 12; higher scores indicate greater symptom severity. The minimally important difference has been defined as a change in total score of greater than 0.3 units. Baseline is mean of 10 days prior to treatment.
Time Frame: Average of 10 days of pre-treatment measurements (day -10 to -1)
Measure: Mean (Standard Deviation); unit: Units on scale, 0-12
Arm/Group | AZD2423 100 mg | Placebo
Number analyzed (Participants) | 31 | 32
Units on scale, 0-12 | 5.2 (1.40) | 5.3 (1.82)

19. Secondary Outcome: BCSS (Evening) Total Score During Last 7 Days of Treatment
Description: The BCSS scale includes one question for each of the symptoms of breathlessness, cough, and sputum. The total BCSS score ranges from 0 to 12; higher scores indicate greater symptom severity. The minimally important difference has been defined as a change in total score of greater than 0.3 units.
Time Frame: Average of the last 7 days of treatment (week 4)
Measure: Mean (Standard Deviation); unit: Units on scale, 0-12
Arm/Group | AZD2423 100 mg | Placebo
Number analyzed (Participants) | 31 | 32
Units on scale, 0-12 | 5.1 (1.68) | 5.1 (2.25)

20. Secondary Outcome: Rescue Medication Use During the Last 7 Days of Treatment
Description: Number of inhalations of short acting β2 agonist (SABA) or short acting muscarinic antagonist (SAMA) per day.
Time Frame: Average of the last 7 days of treatment (week 4)
Measure: Mean (Full Range); unit: Inhalations
Arm/Group | AZD2423 100 mg | Placebo
Number analyzed (Participants) | 30 | 29
Inhalations | 4.0 (1.0) [1.0 to 19.3] | 3.5 (1.0) [1.0 to 7.9]

21. Secondary Outcome: St George's Respiratory Questionnaire for COPD (SGRQ) Total Score at Baseline
Description: The SGRQ-C includes 40 questions in 3 domains: Symptoms (distress due to respiratory symptoms, 7 questions), Activity (disturbance of physical activity, 13 questions), Impacts (overall impact on daily life and well-being, 20 questions). Scores are expressed as a percentage. Baseline is Day 1.
Time Frame: Day 1
Measure: Mean (Standard Deviation); unit: Percent of maximum possible score
Arm/Group | AZD2423 100 mg | Placebo
Number analyzed (Participants) | 31 | 32
Percent of maximum possible score | 55.9 (14.96) | 57.0 (19.27)

22. Secondary Outcome: SGRQ Total Score at End of Treatment
Description: Decrease in score represents improved Quality of Life; increase represents deteriorated Quality of Life. An increase or decrease of 4 or more percent units is judged as the Minimal Clinically Important Difference.
Time Frame: week 4
Measure: Mean (Standard Deviation); unit: Percent of maximum possible score
Arm/Group | AZD2423 100 mg | Placebo
Number analyzed (Participants) | 31 | 32
Percent of maximum possible score | 52.0 (14.38) | 52.9 (18.04)

23. Secondary Outcome: CCL2 (Chemokine Ligand for CCR2b Receptor) Concentration in Plasma at Baseline
Description: Baseline = Day 1 = Visit 2
Time Frame: Day 1
Measure: Geometric Mean (Full Range); unit: pg/mL
Arm/Group | AZD2423 100 mg | Placebo
Number analyzed (Participants) | 29 | 32
pg/mL | 294 [83 to 530] | 279 [111 to 635]

24. Secondary Outcome: CCL2 Concentration in Plasma at End of Treatment
Description: End of treatment = 4 weeks = Visit 6
Time Frame: week 4
Measure: Geometric Mean (Full Range); unit: pg/mL
Arm/Group | AZD2423 100 mg | Placebo
Number analyzed (Participants) | 31 | 32
pg/mL | 1286 [297 to 2410] | 272 [97 to 543]

25. Secondary Outcome: Serum Amyloid-A (SAA) Concentration in Plasma at Baseline
Description: Baseline = Day 1 = Visit 2
Time Frame: Day 1
Measure: Geometric Mean (Full Range); unit: ng/mL
Arm/Group | AZD2423 100 mg | Placebo
Number analyzed (Participants) | 31 | 32
ng/mL | 5175 [964 to 54100] | 4044 [376 to 18600]

26. Secondary Outcome: SAA Concentration in Plasma at End of Treatment
Description: End of treatment = 4 weeks = Visit 6
Time Frame: week 4
Measure: Geometric Mean (Full Range); unit: ng/mL
Arm/Group | AZD2423 100 mg | Placebo
Number analyzed (Participants) | 31 | 32
ng/mL | 6325 [671 to 115000] | 4032 [211 to 320000]

27. Secondary Outcome: Areaa Under the Curve From 0 to 24 Hours (AUC 0-24), Population Pharmacokinetic Evaluation of AZD2423 at Steady State
Description: PK-model: 1-compartment population model with first order absorption. AUC was estimated at steady state
Time Frame: 2 blood samples (pre- and post dose) per visit collected at weeks 1, 2 and 4
Measure: Geometric Mean (Full Range); unit: nmol*h/L
Arm/Group | AZD2423 100 mg | Placebo
Number analyzed (Participants) | 31 | 0
nmol*h/L | 2780 [1370 to 5410] |

28. Secondary Outcome: Cmax, Population Pharmacokinetic Evaluation of AZD2423 at Steady State
Description: PK-model: 1-compartment population model with first order absorption. Cmaxwas estimated at steady state
Time Frame: 2 blood samples (pre- and post dose) per visit collected at weeks 1, 2 and 4
Measure: Geometric Mean (Full Range); unit: nmol/L
Arm/Group | AZD2423 100 mg | Placebo
Number analyzed (Participants) | 31 | 0
nmol/L | 198 [90.7 to 442] |

29. Secondary Outcome: Time to Reach Maximum Concentration (Tmax) Population Pharmacokinetic Evaluation of AZD2423 at Steady State
Description: PK-model: 1-compartment population model with first order absorption. tmax was estimated at steady state
Time Frame: 2 blood samples (pre- and post dose) per visit collected at weeks 1, 2 and 4
Measure: Median (Full Range); unit: Hours
Arm/Group | AZD2423 100 mg | Placebo
Number analyzed (Participants) | 31 | 0
Hours | 1.01 [0.82 to 1.06] |

30. Secondary Outcome: Apparent Volume of Distribution at Steady State (Vss/F) Population Pharmacokinetic Evaluation of AZD2423 at Steady State
Description: PK-model: 1-compartment population model with first order absorption. (Vss/F) was estimated at steady state
Time Frame: 2 blood samples (pre- and post dose) per visit collected at weeks 1, 2 and 4
Measure: Geometric Mean (Full Range); unit: L
Arm/Group | AZD2423 100 mg | Placebo
Number analyzed (Participants) | 31 | 0
L | 1600 [602 to 3650] |

ADVERSE EVENTS:
Arm/Group | AZD2423 100 mg | Placebo
Serious Adverse Events (participants affected / at risk) | 2/31 | 0/32
Other Adverse Events (participants affected / at risk) | 6/31 | 2/32
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | AZD2423 100 mg (N=31) | Placebo (N=32)
Atrial Fibrillation (Cardiac disorders) | 1 (1) | 0 (0)
Atrial Flutter (Cardiac disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | AZD2423 100 mg (N=31) | Placebo (N=32)
Dry Mouth (Gastrointestinal disorders) | 2 | 1
Nasopharyngitis (Infections and infestations) | 2 | 0
Headache (Nervous system disorders) | 2 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Institutions or Investigators were permitted to publish or present the study results from their site (or the overall results), providing the article or presentation was submitted to and approved by AstraZeneca beforehand.